CLINICAL TRIAL: NCT03467776
Title: Brochial Dilation Test by Salbutamol Metered Dose Inhaler(MDI) With Spacer in Wheezy Infants With Asthma Risk Factors
Brief Title: Bronchial Dilation Test in Wheezy Infants
Status: Suspended | Type: Observational
Why Stopped: have to adjust recuriting paticipants projects and have to halted the research
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Firestone Institute for Respiratory Health (Other)
Responsible Party: Principal Investigator, Jinping Zheng, Deputy director,GRID, Guangzhou Institute of Respiratory Disease
Other Study IDs: GIRD201535
Record Dates: First submitted 2018-02-14; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Asthma
Keywords: infants; asthma; bronchial dilation test; plethysmography
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- healthy: healthy control, 5 months to 3 years
- wheezing with atopy: suspected asthma with wheezing (>3 episodes per year) and atopy
- wheezing without atopy: wheezing without atopy

SUMMARY:
The purpose of the study is to establish the methodology of bronchial dilation test by salbutamol MDI with Spacer in wheezy infants with asthma and to evaluate the effects of atopy on the exacerbation of wheeze in wheezy infants.

DETAILED DESCRIPTION:
After screening,each participant undergo baseline pulmonary function test(Jaeger Master Screen Baby Body, Germany)and post-bronchodilator measurements that performed 10min after 200ug of salbutamol administered using a metered-dose inhaler and a spacer.

The participants undergo baseline lung function test and bronchial dilation tests on the second and third visits with one-month interval,and whenever there is an exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* normal term infants.Recurrent wheezing with or without atopy,none of the subjects had a history of respiratory illness, congenital heart disease,dysphagia,oxygen saturation≤90% on room air,an active seizure disorder,or upper airway obstruction,or requirement for assisted ventilation in the neonatal periods,all infants were asymptomatic for at least 2 weeks preceding the test.

Exclusion Criteria:

* subjects had a history of respiratory illness, congenital heart disease,dysphagia,oxygen saturation≤90% on room air,an active seizure disorder,or upper airway obstruction,;all infants were asymptomatic for at least 2 weeks preceding the test.

Ages: 5 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: all the subjects will be recurited from the First Affiliated Hospital of Guangzhou Medical University
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
airway resistance(Raw) performed by body plethysmography before and after bronchial dilation test. | Change from baseline at 20 mins after inhalation of salbutamol
  airway resistance(Raw) at rest

SECONDARY OUTCOMES:
airway resistance(Raw) performed by body plethysmography | at 24 hours of the exacerbation of wheeze
  airway resistance(Raw) measured within 24 hours whenever there is an exacerbation of wheeze.

CONTACTS AND LOCATIONS:
Overall Officials: jinping Zheng, Principal Investigator — Guangzhou Institute of Respiratory Disease
Locations (1):
- State Key Laboratory of Respiratory Disease;China Clinical Research Center of Respiratory Disease;First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No